CLINICAL TRIAL: NCT01904604
Title: Epicutaneous Immunotherapy (EPIT) for Peanut Allergy: A Randomized, Double-Blind, Placebo-Controlled, Phase II Study in Children and Adults (DAIT COFAR6)
Brief Title: Peanut Epicutaneous Phase II Immunotherapy Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Consortium of Food Allergy Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT CoFAR6; 5U19AI066738-07 (NIH)
Record Dates: First submitted 2013-07-15; First posted 2013-07-22 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Peanut Hypersensitivity; Food Hypersensitivity; Hypersensitivity; Hypersensitivity, Immediate
Keywords: Peanut Allergy; Food Allergy; Viaskin peanut patch; Allergen Immunotherapy; Epicutaneous Immunotherapy; Whole peanut extract; Allergenic product; Immediate hypersensitivity
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity; Hypersensitivity; Hypersensitivity, Immediate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Patch (Placebo Comparator): Subjects apply placebo Viaskin® patch daily for a 52-week blinded period. Patch application duration is initially 3 hours and gradually increased to 24 hours over a 21-day graduated dosing period; subsequently patch changed every 24 hours. At Week 52, subjects complete an oral food challenge (OFC) and are unblinded. Following blinded phase, subjects who have not demonstrated sustained unresponsiveness at the Week 52 OFC crossover to active treatment (using the same 21-day graduated dosing period used in the blinded phase) and dose with a high-dose DBV712 Viaskin® patch containing 250 μg peanut protein for a total active treatment period of 30 months (130 weeks).
  Interventions: Biological: Placebo Viaskin® Patch
- 100 µg Peanut Patch (Experimental): Subjects apply low-dose DBV712 Viaskin® patch containing 100 micrograms (μg) peanut protein daily for a 52-week blinded period. Patch application duration is initially 3 hours and gradually increased to 24 hours over a 21-day graduated dosing period; subsequently patch changed every 24 hours. At Week 52, subjects complete an OFC and are unblinded. Following blinded phase, subjects who have not demonstrated sustained unresponsiveness at the Week 52 OFC crossover to active treatment (using same 21-day graduated dosing period used in blinded phase for subjects 4-<6 years old at enrollment or who had Grade 2 reaction or higher within previous 2 months) and dose with a high-dose DBV712 Viaskin® patch containing 250 μg peanut protein for a total active treatment period of 30 months (130 weeks).
  Interventions: Biological: Low-dose DBV712 Viaskin® Patch
- 250 µg Peanut Patch (Experimental): Subjects apply high-dose DBV712 Viaskin® patch containing 250 micrograms (μg) peanut protein daily for a 52-week blinded period. Patch application duration is initially 3 hours and gradually increased to 24 hours over a 21-day graduated dosing period; subsequently patch changed every 24 hours. At Week 52, subjects complete an OFC and are unblinded. Following blinded phase, subjects who have not demonstrated sustained unresponsiveness at the Week 52 OFC continue active treatment with a high-dose DBV712 Viaskin® patch for a total active treatment period of 30 months (130 weeks).
  Interventions: Biological: High-dose DBV712 Viaskin® Patch

INTERVENTIONS:
Biological: Placebo Viaskin® Patch — Placebo (e.g., no peanut) patch in an epicutaneous application for 24 hours every 24 hours.
  Arms: Placebo Patch
Biological: Low-dose DBV712 Viaskin® Patch — 100 microgram (µg) dose of peanut proteins in an epicutaneous application for 24 hours every 24 hours.
  Arms: 100 µg Peanut Patch
Biological: High-dose DBV712 Viaskin® Patch — 250 microgram (µg) dose of peanut proteins in an epicutaneous application for 24 hours every 24 hours.
  Arms: 250 µg Peanut Patch

SUMMARY:
Food allergy occurs when the immune system reacts against foods. The immune system is the part of the body that protects us from illness and germs, but it can also cause allergies. Peanut allergy occurs in 1 - 2% of people in the United States and other Western countries. There is proof that allergy to peanut is increasing. Allergic reactions to peanut can be severe and life threatening. The only way that you can prevent an allergic reaction is to avoid exposure to peanuts. However, peanut proteins are found in a variety of foods and people can be accidently exposed to peanut proteins. Treatment for accidental exposure include antihistamines (medications like Benadryl), and injectable epinephrine (adrenalin) which must be carried at all times. DBV Technologies has developed an epicutaneous delivery system, a patch that puts the peanut protein on the skin.

DETAILED DESCRIPTION:
This study will evaluate whether peanut epicutaneous immunotherapy can protect individuals who are allergic to peanuts from having severe allergic reactions, when accidentally exposed to peanuts. The study also looks at the safety of the treatment and the effects it has on the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed peanut allergy OR convincing history of peanut allergy
* A skin prick test positive to peanut (wheal diameter ≥3mm greater than the saline control) OR detectable peanut specific Immunoglobulin E (IgE) (ImmunoCAP >0.35 kUA/L)
* Positive reaction to a cumulative dose of ≤1044 mg peanut protein in the initial qualifying Oral Food Challenge (OFC)
* Use of an effective method of contraception by females of childbearing potential to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of their participation in the study
* Ability to perform spirometry maneuvers in accordance with the American Thoracic Society (ATS) guidelines (1994). Children ages 4-11 years who have documented inability to adequately perform spirometry may be enrolled if Peak Expiratory Flow (PEF) is >80% of predicted
* Provide signed informed consent or assent where indicated

Exclusion Criteria:

* History of anaphylaxis to peanut resulting in hypotension, neurological compromise or requiring mechanical ventilation
* Participation in a study using an investigational new drug in the last 30 days
* Participation in any interventional study for the treatment of food allergy in the past 6 months
* Pregnancy or lactation
* Current or known allergy to the Viaskin Peanut/Placebo patch device or excipients
* Current or known allergy to the placebo allergen (oat flour) in oral food challenge (OFC)
* Currently in a build-up phase of any allergen immunotherapy
* Severe or poorly controlled atopic dermatitis or greater than a mild flare of active disease at enrollment
* Forced Expiratory Volume in 1 Second (FEV1) value <80% predicted or any clinical features of moderate or severe persistent asthma baseline severity (as defined by the 2007 NHLBI Guidelines) and greater than high daily doses of inhaled corticosteroids (>500mcg of Fluticasone or equivalent)
* Use of steroid medications in the following manners: history of daily oral steroid dosing for >1 month during the past year, or burst or steroid course in the past 3 months, or >1 burst oral steroid course in the past year or use of oral or parenteral steroids for a non-asthma indication within the past 30 days
* Asthma requiring >1 hospitalization in the past year for asthma or >1 Emergency Department (ED) visit in the past 6 months for asthma
* Any previous intubation/mechanical ventilation due to allergies or asthma
* Use of omalizumab or other non-traditional forms of allergen immunotherapy or immunomodulatory or biologic therapy in the past year
* Use of beta-adrenergic blockers, angiotensin-converting enzyme inhibitors, angiotensin-receptor blockers, or calcium channel blockers in the past 30 days
* Inability to discontinue antihistamines for skin testing and OFC
* History of alcohol or drug abuse
* History of cardiovascular disease, uncontrolled hypertension, arrhythmias, chronic lung disease, active eosinophilic gastrointestinal disease, or other medical conditions including immunologic disorders or HIV infection which, in the opinion of the investigator, make the subject unsuitable for treatment or at increased risk of anaphylaxis or poor outcome

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2018-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacie M. Jones, MD, Study Chair — University of Arkansas
Locations (5):
- United States (5):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - National Jewish Health, Denver, Colorado
  - The Johns Hopkins University, Baltimore, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill School of Medicine, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data in ImmPort [https://immport.niaid.nih.gov/ ], a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: After completion of the trial.
Access Criteria: After completion of the trial.
URL: https://immport.niaid.nih.gov/

REFERENCES:
- [Background] Keet CA, Wood RA. Emerging therapies for food allergy. J Clin Invest. 2014 May;124(5):1880-6. doi: 10.1172/JCI72061. Epub 2014 May 1. PMID 24789880
- [Result] Jones SM, Sicherer SH, Burks AW, Leung DY, Lindblad RW, Dawson P, Henning AK, Berin MC, Chiang D, Vickery BP, Pesek RD, Cho CB, Davidson WF, Plaut M, Sampson HA, Wood RA; Consortium of Food Allergy Research. Epicutaneous immunotherapy for the treatment of peanut allergy in children and young adults. J Allergy Clin Immunol. 2017 Apr;139(4):1242-1252.e9. doi: 10.1016/j.jaci.2016.08.017. Epub 2016 Oct 26. PMID 28091362
- [Derived] Scurlock AM, Burks AW, Sicherer SH, Leung DYM, Kim EH, Henning AK, Dawson P, Lindblad RW, Berin MC, Cho CB, Davidson WF, Plaut M, Sampson HA, Wood RA, Jones SM; Consortium for Food Allergy Research (CoFAR). Epicutaneous immunotherapy for treatment of peanut allergy: Follow-up from the Consortium for Food Allergy Research. J Allergy Clin Immunol. 2021 Mar;147(3):992-1003.e5. doi: 10.1016/j.jaci.2020.11.027. Epub 2020 Dec 5. PMID 33290772
- [Derived] Chiang D, Chen X, Jones SM, Wood RA, Sicherer SH, Burks AW, Leung DYM, Agashe C, Grishin A, Dawson P, Davidson WF, Newman L, Sebra R, Merad M, Sampson HA, Losic B, Berin MC. Single-cell profiling of peanut-responsive T cells in patients with peanut allergy reveals heterogeneous effector TH2 subsets. J Allergy Clin Immunol. 2018 Jun;141(6):2107-2120. doi: 10.1016/j.jaci.2017.11.060. Epub 2018 Jan 31. PMID 29408715
- See also: National Institute of Allergy and Infectious Diseases (NIAID) Website — https://www.niaid.nih.gov/
- See also: Consortium of Food Allergy Research (CoFAR) Website — http://www.cofargroup.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from September 2013 to July 2014 at the five listed university-based medical centers located in the United States.
Period: Overall Study
Arm/Group | Placebo Patch | 100 µg Peanut Patch | 250 µg Peanut Patch
Started | 25 | 25 | 25
Completed Week 52 OFC (Completion of the Week 52 OFC was required to assess the primary endpoint of the study.) | 22 | 21 | 25
Began Crossover Treatment | 20 (2 participants who completed the Week 52 OFC did not crossover; 1 passed the OFC and 1 relocated.) | 21 | 0 (Per protocol, this treatment group did not crossover.)
Completed Week 130 OFC | 18 | 18 | 23
Completed | 18 (COMPLETED: Completed the Week 130 Oral Food Challenge (OFC).) | 18 (COMPLETED: Completed the Week 130 Oral Food Challenge (OFC).) | 23 (COMPLETED: Completed the Week 130 Oral Food Challenge (OFC).)
Not Completed | 7 | 7 | 2
Not completed — Withdrew before receiving dosing | 0 | 1 | 0
Not completed — Non-compliance | 1 | 0 | 0
Not completed — Anxiety about OFC/Refused OFC | 2 | 0 | 0
Not completed — Patch site reactions | 1 | 1 | 0
Not completed — Increased syncope | 0 | 1 | 0
Not completed — Unrelated illness | 0 | 1 | 0
Not completed — Passed Week 52 OFC | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Participant Relocated | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects who received study treatment. Note that 1 subject in the 100 µg Peanut Patch group who never received treatment was not included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Patch | 100 µg Peanut Patch | 250 µg Peanut Patch | Total
Number analyzed (Participants) | 25 | 24 | 25 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 24 | 25 | 73
  Between 18 and 65 years | 1 | 0 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (3.9) | 9.7 (3.4) | 8.8 (3.4) | 9.5 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 9 | 28
  Male | 16 | 14 | 16 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 4
  Not Hispanic or Latino | 24 | 24 | 22 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3
  White | 22 | 18 | 23 | 63
  More than one race | 0 | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 25 | 74
Atopic Dermatitis Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The Atopic Dermatitis Total Score is scored on a 10 point scale of 0 to 9 where a higher score indicates increasing severity of atopic dermatitis. This score is a combination of three scores that range from 0 to 3 in the following areas: body surface area score, disease course, and disease intensity.
  Scores on a scale | 1.9 (2.6) | 1.4 (2.3) | 1.5 (2.2) | 1.6 (2.4)
Total IgE [Mean (Standard Deviation); unit: kU/L] — Total amount of serum immunoglobulin E.
  kU/L | 751.8 (797.6) | 949.1 (1183.5) | 691.5 (602.3) | 795.4 (884.2)
Peanut IgE [Mean (Standard Deviation); unit: kUA/L] — Amount of serum peanut-specific immunoglobulin E. Individuals with a peanut IgE of <0.35 kUA/L are considered not to be sensitized to peanut.
  kUA/L | 77.3 (69.4) | 87.6 (65.3) | 89.9 (64.3) | 84.9 (65.7)
Skin Prick Test Score [Mean (Standard Deviation); unit: mm] — This score is calculated by subtracting the size of the saline wheal (in mm) from the size of the peanut wheal (in mm) observed for a skin prick test. Individuals with a peanut skin prick test score of < 3 mm are considered to have a negative result.
  mm | 14.1 (8.6) | 12.9 (6.8) | 12.7 (5.2) | 13.3 (7.0)
Age at Initial Peanut Allergic Reaction [Mean (Standard Deviation); unit: years] | 1.9 (1.2) | 2.8 (3.3) | 2.1 (2.0) | 2.3 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a Successful Treatment Response
Description: Treatment response is defined as a subject who can either (a) successfully consume a cumulative dose of peanut protein equal to or greater than 5044 mg or (b) successfully consume at least a 10-fold increase in peanut protein at the Week 52 oral food challenge (OFC), when compared to the cumulative successfully consumed dose at the baseline OFC.
Time Frame: Week 52
Population: All randomized subjects who received study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Patch | 100 µg Peanut Patch | 250 µg Peanut Patch
Number analyzed (Participants) | 25 | 24 | 25
percentage of participants | 12.0 | 45.8 | 48.0
Statistical Analysis 1: Comparison: Placebo Patch vs 100 µg Peanut Patch; The null hypothesis was that there was no difference between treatment groups. Subjects who did not complete the Week 52 oral food challenge were counted as treatment failures; Test type: Superiority or Other; p = 0.005, Barnard's statistic — A one-sided test was used with the a priori threshold for statistical significance of 0.0125. No adjustments were made to the p-value; Risk Difference (RD) = 33.8, 33.8% CI 2-sided [10.2 to 57.5]
Statistical Analysis 2: Comparison: Placebo Patch vs 250 µg Peanut Patch; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.003, Barnard's statistic — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 36.0, 36.0% CI 2-sided [12.6 to 59.4]
Statistical Analysis 3: Comparison: 100 µg Peanut Patch vs 250 µg Peanut Patch; Test type: Superiority or Other; p = 0.48, Barnard's statistic — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 2.2, 2.2% CI 2-sided [-25.8 to 30.1]

2. Secondary Outcome: Percentage of Subjects Desensitized to Peanut Protein
Description: Desensitization is defined based on successfully consumed dose in mg protein at the Week 130 oral food challenge (OFC) as follows:
  1) 0-44 mg at BL, >=444 mg at Wk 130 2) >44-<444 mg at BL, 10-fold increase at Wk 130 3) >=444 mg at BL, >=5,044 mg at Wk 130.
  BL=Baseline, Wk 130=Week 130 (Month 30)
Time Frame: Week 130 (Month 30)
Population: All randomized subjects who received active (not placebo) study treatment. For the Placebo Patch group, this only includes the 20 subjects who crossed over to active treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Patch | 100 µg Peanut Patch | 250 µg Peanut Patch
Number analyzed (Participants) | 20 | 24 | 25
percentage of participants | 5.0 [0.1 to 24.9] | 20.8 [7.1 to 42.2] | 36.0 [18.0 to 57.5]

3. Secondary Outcome: Percentage of Subjects Who Can Successfully Consume 1044 mg or 5044 mg Peanut Protein
Description: Subjects who successfully consumed without dose-limiting symptoms 1044 mg or 5044 mg peanut protein during the Week 130 oral food challenge (OFC). This is referred to as the successfully consumed dose (SCD). The maximum SCD for this OFC was 5044 mg peanut protein.
Time Frame: Week 130 (Month 30)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Patch | 100 µg Peanut Patch | 250 µg Peanut Patch
Number analyzed (Participants) | 20 | 24 | 25
percentage of participants
  SCD>=1044 mg peanut protein | 10.0 [1.2 to 31.7] | 16.7 [4.7 to 37.4] | 32.0 [14.9 to 53.5]
  SCD=5044 mg peanut protein | 0.0 [0.0 to 16.8] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 13.7]

4. Secondary Outcome: Percentage of Desensitized Subjects in the Active Treatment Arms as Measured by 5044 mg Peanut Protein Oral Food Challenge (OFC)
Description: Desensitization is defined based on successfully consumed dose in mg protein at the Week 52 oral food challenge (OFC) as follows:
  0-44 mg at BL, >=444 mg at Wk52 2) >44-<444 mg at BL, 10-fold increase at Wk 52 3) >=444 mg at BL, >=5,044 mg at Wk 52.
  BL=Baseline, Wk 52=Week 52
Time Frame: Week 52
Population: All randomized subjects who received active (not placebo) study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | 100 µg Peanut Patch | 250 µg Peanut Patch
Number analyzed (Participants) | 24 | 25
percentage of participants | 12.5 | 20.0

5. Secondary Outcome: Average Successfully Consumed Dose as Measured by 5044 mg Peanut Protein Oral Food Challenge (OFC)
Description: The successfully consumed dose (SCD) is the cumulative dose consumed during an oral food challenge without dose-limiting symptoms that led to the termination of the challenge.
Time Frame: Week 52
Population: All randomized subjects who completed the Week 52 OFC.
Measure: Median (Full Range); unit: mg protein
Arm/Group | Placebo Patch | 100 µg Peanut Patch | 250 µg Peanut Patch
Number analyzed (Participants) | 22 | 21 | 25
mg protein | 14 [1 to 5044] | 144 [44 to 2044] | 144 [0 to 2044]
Statistical Analysis 1: Comparison: 100 µg Peanut Patch vs 250 µg Peanut Patch; The null hypothesis was that there was no difference between treatment groups; Test type: Superiority or Other; p = 0.80, Wilcoxon (Mann-Whitney) — No adjustments were made to the p-value; The two-sided t approximation was used
Statistical Analysis 2: Comparison: Placebo Patch vs 100 µg Peanut Patch; The null hypothesis was that there was no difference between treatment groups; Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney) — No adjustments were made to the p-value; The two-sided t approximation was used
Statistical Analysis 3: Comparison: Placebo Patch vs 250 µg Peanut Patch; The null hypothesis was that there was no difference between treatment groups; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney) — No adjustments were made to the p-value; The two-sided t approximation was used

6. Secondary Outcome: Percentage of Subjects Who Pass an OFC to 5044 mg of Peanut Protein Followed by an Open Feeding of Peanut Butter After 8 Weeks or 20 Weeks of Discontinuation of Dosing Subsequent to Passing the Week 130 Oral Food Challenge (OFC)
Description: Subjects who after passing the Week 130 (Month 30) discontinue dosing for 8 weeks and later 20 weeks successfully consumed 5044 mg peanut protein during an OFC followed by an open feeding of peanut butter.
Time Frame: 8 and 20 weeks after the Week 130 (Month 30) OFC
Population: None of the participants passed the Week 130 OFC so this could not be assessed.
Arm/Group | Placebo Patch | 100 µg Peanut Patch | 250 µg Peanut Patch
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Percentage of Subjects With Adverse Events Related to Therapy Through Week 52 and Through 30 Months
Description: Adverse events (AEs) related to study therapy includes both unsolicited AEs where there was a reasonable possibility that the study product caused the event as well as solicited AEs related to dosing.
Time Frame: Week 52 and Month 30 (Week 130)
Population: All randomized subjects who received study treatment were included in the analysis. For the Placebo Patch group, at Week 130 only the 20 participants who crossed over to active treatment were included.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Patch | 100 µg Peanut Patch | 250 µg Peanut Patch
Number analyzed (Participants) | 25 | 24 | 25
percentage of participants
  Had AE related to study therapy through Week 52 | 88.0 | 100.0 | 100.0
  Had AE related to study therapy through Month 30 | 100.0 | 100.0 | 100.0

8. Secondary Outcome: Percentage of Subjects Who Successfully Complete the Dosing Regimen With no More Than Mild Symptoms Related to Peanut Patch Dosing After 30 Months of Therapy
Description: Mild symptoms related to peanut patch dosing are defined as patch site reactions up to Grade 2 in severity or mild systemic dosing symptoms.
Time Frame: Month 30 (Week 130)
Population: All randomized subjects who received active (not placebo) study treatment. The Placebo Patch group includes the 20 subjects who crossed over to active treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Patch | 100 µg Peanut Patch | 250 µg Peanut Patch
Number analyzed (Participants) | 20 | 24 | 25
percentage of participants | 65.0 | 62.5 | 64.0

ADVERSE EVENTS:
Time Frame: For the Placebo Patch group, data were collected for 52 weeks of double-blind dosing with a placebo patch and 130 weeks of open label dosing on active treatment with the DBV712 Viaskin® Patch with 250 µg peanut protein. For the 100 µg Peanut Patch group and the 250 µg Peanut Patch group, data were collected for 52 weeks of double-blind dosing and then 78 weeks of open label dosing for a total of 130 weeks of active treatment.
Description: This study graded the severity of Adverse Events experienced by participants according to the criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.
Groups:
- Placebo Patch Before Week 52 OFC (Double Blind): Subjects apply placebo Viaskin® patch daily for a 52-week blinded period. Patch application duration is initially 3 hours and gradually increased to 24 hours over a 21-day graduated dosing period; subsequently patch changed every 24 hours. At Week 52, subjects complete an oral food challenge (OFC) and are unblinded. Following blinded phase, subjects who have not demonstrated sustained unresponsiveness at the Week 52 OFC crossover to active treatment (using the same 21-day graduated dosing period used in the blinded phase) and dose with a high-dose DBV712 Viaskin® patch containing 250 μg peanut protein for a total active treatment period of 30 months (130 weeks).
  Placebo Viaskin® Patch: Placebo (e.g., no peanut) patch in an epicutaneous application for 24 hours every 24 hours.
- Placebo Patch Crossed Over to 250 µg Peanut Patch (Open Label): After 52 weeks of double-blind Placebo Patch therapy, subjects complete an oral food challenge (OFC) and are unblinded. Following blinded phase, subjects who have not demonstrated sustained unresponsiveness at the Week 52 OFC crossover to active treatment (using the same 21-day graduated dosing period used in the blinded phase) and dose with a high-dose DBV712 Viaskin® patch containing 250 μg peanut protein for a total active treatment period of 30 months (130 weeks).
  High-dose DBV712 Viaskin® Patch: 250 microgram (µg) dose of peanut proteins in an epicutaneous application for 24 hours every 24 hours.
Arm/Group | Placebo Patch Before Week 52 OFC (Double Blind) | Placebo Patch Crossed Over to 250 µg Peanut Patch (Open Label) | 100 µg Peanut Patch | 250 µg Peanut Patch
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/20 | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/20 | 2/24 | 0/25
Other Adverse Events (participants affected / at risk) | 23/25 | 20/20 | 24/24 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Patch Before Week 52 OFC (Double Blind) (N=25) | Placebo Patch Crossed Over to 250 µg Peanut Patch (Open Label) (N=20) | 100 µg Peanut Patch (N=24) | 250 µg Peanut Patch (N=25)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Patch Before Week 52 OFC (Double Blind) (N=25) | Placebo Patch Crossed Over to 250 µg Peanut Patch (Open Label) (N=20) | 100 µg Peanut Patch (N=24) | 250 µg Peanut Patch (N=25)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (2) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 4 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (5) | 5 (8)
Application site erythema (General disorders) | 19 (1125) | 20 (13802) | 24 (12823) | 25 (16443)
Application site extravasation (General disorders) | 8 (329) | 19 (5335) | 22 (4822) | 25 (5066)
Application site papules (General disorders) | 6 (128) | 16 (2918) | 23 (2725) | 25 (4575)
Application site pruritus (General disorders) | 18 (728) | 20 (11580) | 24 (9175) | 25 (14214)
Application site reaction (General disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 5 (5) | 4 (7) | 6 (11) | 8 (11)
Allergy to animal (Immune system disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (2)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ear infection (Infections and infestations) | 2 (4) | 2 (4) | 2 (3) | 1 (1)
Gastoenteritis viral (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 4 (4)
Gastroenteritis (Infections and infestations) | 3 (5) | 1 (1) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 4 (4)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Pharyngitis streptococcal (Infections and infestations) | 2 (3) | 2 (2) | 3 (9) | 7 (12)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 8 (14)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 7 (10) | 11 (21) | 15 (26)
Viral infection (Infections and infestations) | 1 (3) | 2 (3) | 3 (3) | 7 (7)
Viral upper respiratory tract infection (Infections and infestations) | 3 (5) | 5 (11) | 5 (9) | 7 (15)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 4 (12) | 3 (10)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 6 (8) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5) | 4 (4) | 4 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (5) | 3 (4) | 5 (7) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (4) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (11) | 4 (6) | 4 (8) | 4 (7)
Mole excision (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 2 (4) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tonsilitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (8) | 1 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No